CLINICAL TRIAL: NCT01329315
Title: Tailored Youth Drug Intervention In Primary Care
Brief Title: Project Chill: Tailored Youth Drug Intervention In Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frederic C. Blow, Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: DA020075; R01DA020075-01 (NIH)
Record Dates: First submitted 2011-03-29; First posted 2011-04-05 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Marijuana Use
MeSH Terms: conditions — Marijuana Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BMI-T (Active Comparator): Brief Motivational Intervention (BMI-T): social worker/therapist-delivered intervention (25-minute tailored structured module).
  Interventions: Behavioral: BMI-T
- BMI-C (Active Comparator): Computer-delivered intervention (BMI-C): computerized tailored 25-minute intervention.
  Interventions: Behavioral: BMI-C
- DPB (No Intervention): Drug Prevention Booklet (DPB)- National Institute on Drug Abuse (NIDA)-developed drug prevention booklet to address preventing marijuana initiation, and marijuana use.

INTERVENTIONS:
Behavioral: BMI-T — Brief Motivational Intervention (BMI-T): social worker/therapist-delivered intervention (25-minute tailored structured module).
  Arms: BMI-T
Behavioral: BMI-C — Computer-delivered intervention (BMI-C): computerized tailored 25-minute intervention.
  Arms: BMI-C

SUMMARY:
This study examines the impact of tailored computer-delivered and therapist-delivered brief motivations prevention/interventions both for adolescents who have not initiated marijuana use (prevention), and those who use marijuana (intervention). Key moderators of prevention/intervention effectiveness will be examined, including behavioral intentions, self-efficacy, stage of change, school involvement, susceptibility to peer pressure, and potential health consequences such as STD/HIV risk behaviors. This project will provide the critical first step toward the development and implementation of marijuana use prevention/intervention programs that have the potential to be delivered to a large segment of youth who seek care in our nation's primary care settings.

DETAILED DESCRIPTION:
The primary care setting represents an underutilized venue for prevention interventions addressing drug use/abuse among youth. The purpose of the study is to: (1) develop and refine promising, empirically-derived, BMI prevention/intervention modules delivered by a clinician or a computer to target marijuana use, and (2) test the effectiveness of BMI in preventing initiation/escalation of marijuana use among youth in community health clinics. This randomized controlled trial screened adolescents in primary care clinics in Flint, MI. A random sample of those who screened negative for past year marijuana use were selected to participate in the study and all subjects who screened positive for past year use were enrolled in the study. These subjects were stratified by gender, age, and past year marijuana use and randomized to one of three conditions: 1) computer-delivered brief motivational approach (BMI-C); 2) therapist-delivered brief motivational approach (BMI-T); or 3) a NIDA drug education booklet. Primary outcomes are evaluated at 3-, 6- and 12-months and include marijuana, alcohol, tobacco and other drug use. Key moderators of effectiveness will be examined, including behavioral intentions, self-efficacy, stage of change, school involvement, susceptibility to peer pressure, and potential health consequences (e.g., STD/HIV risk behaviors). This project will provide the critical first step toward the implementation of tailored marijuana prevention and intervention in primary care clinics.

ELIGIBILITY:
Inclusion Criteria:

* adolescents (ages 12-18) presenting to the approved health clinics (except exclusions as noted below)
* ability to provide informed assent
* access to a parent or guardian for parental consent

Exclusion Criteria:

* adolescents who do not understand English
* adolescents deemed unable to provide informed consent by research staff (e.g., cognitive issues)
* adolescents who come to the clinic because of sexual assault or suicide attempt, or are presenting with high psychological distress requiring intensive attention
* prisoners
* adolescents who are deaf
* adolescents with a sibling or other household member in the study will be excluded from Phase II

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1141 (Actual)
Dates: Start 2005-09; Primary Completion 2010-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
marijuana use | 12 months
  initiation of marijuana use or escalation of use

SECONDARY OUTCOMES:
alcohol, tobacco, and illicit drug use | 12 months
  initiation of drug use (defined as tobacco, alcohol, marijuana, or other drugs), escalation of substance use within substances (e.g., increased frequency of use), escalation of drug use to other substances (movement from tobacco to alcohol, or alcohol to marijuana, or marijuana to other "harder" drugs
risk involvement | 12 months
  delinquency, peer affiliation and social context influences

CONTACTS AND LOCATIONS:
Overall Officials: Frederic C Blow, PhD, Principal Investigator — University of Michigan

REFERENCES:
- [Derived] Walton MA, Bohnert K, Resko S, Barry KL, Chermack ST, Zucker RA, Zimmerman MA, Booth BM, Blow FC. Computer and therapist based brief interventions among cannabis-using adolescents presenting to primary care: one year outcomes. Drug Alcohol Depend. 2013 Oct 1;132(3):646-53. doi: 10.1016/j.drugalcdep.2013.04.020. Epub 2013 May 25. PMID 23711998